CLINICAL TRIAL: NCT01645085
Title: An Open-label, Single-center, Randomized, 4-way Crossover Study to Assess the Bioequivalence of R406 in Healthy Volunteers When 100 and 150mg of Fostamatinib Are Administered as the 13% Drug-loaded Tablet Versus the 38% Drug-loaded Tablet
Brief Title: A Study to Assess the Bioequivalence of R406 in Healthy Volunteers When Given 100mg and 150 mg of Fostamatinib
Acronym: Fosta BE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00020
Record Dates: First submitted 2012-07-13; First posted 2012-07-20 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Volunteers
Keywords: R406; Fostamatinib; Phase I; Healthy Subjects; Pharmacokinetics; Bioequivalence

ARMS (4):
- Treatment A (Experimental): 100mg MCC-based 13% drug-loaded tablets
  Interventions: Drug: MCC-based 13% drug loaded tablets
- Treatment B (Experimental): 100mg mannitol-based 38% drug-loaded tablets
  Interventions: Drug: Mannitol-based 38% drug-loaded tablet
- Treatment C (Experimental): 150mg MCC-based 13% drug-loaded tablets
  Interventions: Drug: MCC-based 13% drug loaded tablets
- Treatment D (Experimental): 150mg mannitol-based 38% drug-loaded tablets
  Interventions: Drug: Mannitol-based 38% drug-loaded tablet

INTERVENTIONS:
Drug: MCC-based 13% drug loaded tablets — 50mg tablets, dosed as 2 tablets (100mg total)
  Arms: Treatment A
Drug: Mannitol-based 38% drug-loaded tablet — One 100mg tablet
  Arms: Treatment B
Drug: MCC-based 13% drug loaded tablets — 3 tablets (150mg total)
  Arms: Treatment C
Drug: Mannitol-based 38% drug-loaded tablet — One 150 mg tablet
  Arms: Treatment D

SUMMARY:
A study in Healthy Volunteers to Compare the Amount of R406 in Blood When Given Different Formulations of Fostamatinib.

DETAILED DESCRIPTION:
An Open-label, Single-center, Randomized, 4-way Crossover Study to Assess the Bioequivalence of R406 in Healthy Volunteers when 100 and 150mg of Fostamatinib are Administered as the 13% Drug-loaded Tablet Versus the 38% Drug-loaded Tablet.

Treatment sequences will be determined using two 2-2 crossover designs in sequence, 1 for treatments A and B, and 1 for treatments C and D. The order of the designs containing AB/BA and CD/DC within the overall design, as well as the order of treatments within each design, will be randomized. This gives a total of 8 possible treatment sequences as follows: ABCD, ABDC, BACD, BADC, CDAB, CDBA, DCAB, DCBA.

ELIGIBILITY:
Inclusion Criteria:

* Males and nonlactating, non childbearing potential females from 18 to 55 years, inclusive and with a weight of at least 50 kg and BMI between 18 and 30 kg/m2, inclusive
* Females must have a negative pregnancy test at screening and on admission to the study center of each period, must not be lactating and must be of non childbearing potential
* Non childbearing potential can be confirmed by being postmenopausal defined as amenorrhea for a least 12 months following cessation of all exogenous hormonal treatments and with FSH and LH levels in the laboratory-defined postmenopausal range
* Non childbearing potential can be confirmed by documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation.

Exclusion Criteria:

* History of any clinically significant disease or disorder, including GI, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody
* Known or suspected history of drug abuse, as judge by the investigator
* Any clinically significant abnormalities on 12-lead ECG as judged by the Investigator
* Current smokers, or those who have smoked, used nicotine-containing products, or used smoking cessation treatments within the previous 1 month prior to enrollment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence of R406 when fostamatinib is administered as two 50mg MCC-based 13% drug-loaded tablets versus one 100mg mannitol-based 38% drug-loaded tablet | Measured at predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours postdose
Bioequivalence of R406 when fostamatinib is administered as three 50mg MCC-based 13% drug-loaded tablets versus one 150mg mannitol-based 38% drug-loaded tablet | Measured at predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours postdose

SECONDARY OUTCOMES:
AUC for mannitol-based 38% drug-loaded tablets and MCC-based 13% drug-loaded tablets | Measured at predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours postdose
Cmax for mannitol-based 38% drug-loaded tablets and MCC-based 13% drug-loaded tablets | Measured at predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours postdoses
Frequency of adverse events | Measured throughout the study and 3 -5 days after discharge from Period 4, approximately 45 days
Severity of adverse events | Measured throughout the study and 3 -5 days after discharge from Period 4, approximately 45 days

CONTACTS AND LOCATIONS:
Overall Officials: Chris O'Brien, MEDICAL SCIENCE DIRECTOR, Study Director — AstraZeneca; David Mathews, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Overland Park, Kansas, United States